CLINICAL TRIAL: NCT02350946
Title: Effects of Oxytocin on Emotion Recognition and Response Inhibition
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EK163/13
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: The Impact of Oxytocin on Social Cognition
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cross over Oxytocin and Placebo (Experimental): fMRI measurement and blood examinations following 26 IU Oxytocin (Syntocinon) on day 1 and following placebo on day 14
  Interventions: Drug: Oxytocin; Drug: Placebo
- Cross over Placebo and Oxytocin (Experimental): fMRI measurement and blood examinations following placebo on day 1 and following 26 IU Oxytocin (Syntocinon) on day 14
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
Drug: Placebo

SUMMARY:
The purpose of this study is to shed light on the basic neurobiological mechanisms which underlie social information processing in healthy men. More specifically, we intend to examine whether a person's social competence level is related to the patterns of neural activity and his visual search strategies during evaluation of social scenes. Furthermore, it will be assessed whether an oxytocin-driven increase in activity in brain areas relevant to the task will facilitate social information processing and thus enhance task performance. Additionally it will be examined whether oxytocin can facilitate response inhibition in an emotional context.

ELIGIBILITY:
Inclusion Criteria:

* MRI- eligibility
* Subject's ability to fully grasp the type, scope and individual consequences of the study
* Willingness to participate in and comply with the study procedures as indicated by signing the dated informed consent form

Exclusion Criteria:

* Left-handedness
* Smoking
* Regular intake of medication
* Hypersensitivity towards oxytocin or a chemically similar substance
* Current or previous neurological or psychiatric disorder
* Nose surgery or chronic sinus infection
* Any somatic disorder that may interfere with the experimental procedures, affect the outcome measures or pose a risk for the participant during performance of the experiment

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
BOLD response during emotion recognition in contrast with a corresponding control condition. | (Day 1: oxytocin, Day: 14:placebo, or vice versa [counterbalanced])
  In the Social Detection Task, subjects' brain activity when viewing social scenes will be compared to corresponding control scenes in which no people are shown.
  In the GoNoGo Task several emotional conditions will be compared to a neutral control condition.
BOLD response during response inhibition (Emotional Go/ Nogo) in contrast with a corresponding control condition. | (Day 1: oxytocin, Day: 14:placebo, or vice versa [counterbalanced])
  Brain activation during NoGo trials will be compared to brain activation during Go trials from the same emotional condition.

SECONDARY OUTCOMES:
Serum levels of Oxytocin | (Day 1: oxytocin, Day: 14:placebo, or vice versa [counterbalanced])
Serum levels of Prolaktin | (Day 1: oxytocin, Day: 14:placebo, or vice versa [counterbalanced])
Serum levels of Cortisol | (Day 1: oxytocin, Day: 14:placebo, or vice versa [counterbalanced])
Total length of fixations on areas of interest (AOIs) assessed via eye-tracking | (Day 1: oxytocin, Day: 14:placebo, or vice versa [counterbalanced])
  In the SoDeTa stimulus set, faces, arms and hands were defined as 1st order AOIs and remaining parts of the body as 2nd order AOIs.
  In the GoNoGo task, for each stimulus, the eye region of the face was chosen as AOI.
Number of fixations on areas of interest (AOIs) assessed via eye-tracking | (Day 1: oxytocin, Day: 14:placebo, or vice versa [counterbalanced])
  In the SoDeTa stimulus set, faces, arms and hands were defined as 1st order AOIs and remaining parts of the body as 2nd order AOIs.
  In the GoNoGo task, for each stimulus, the eye region of the face was chosen as AOI.
Percentage of correct responses in an emotion recognition paradigm (Social Detection Task) and a response inhibition task (Emotional Go/Nogo). | (Day 1: oxytocin, Day: 14:placebo, or vice versa [counterbalanced])
Response time in an emotion recognition paradigm (Social Detection Task) and a response inhibition task (Emotional Go/Nogo). | (Day 1: oxytocin, Day: 14:placebo, or vice versa [counterbalanced])

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital RWTH Aachen, Aachen, Germany